CLINICAL TRIAL: NCT05344989
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of APNmAb005 in Healthy Subjects
Brief Title: A First-in-Human Study to Assess Single Doses of APNmAb005 in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: APRINOIA Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Organization: APRINOIA Therapeutics (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APNmAb005-101
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers; Tauopathies; Alzheimer Disease
Keywords: Healthy Volunteers; Alzheimer's Disease; Alzheimer Disease; AD; Tauopathies; Tau
MeSH Terms: conditions — Tauopathies; Alzheimer Disease; Pick Disease of the Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- APNmAb005 (5mg/kg) vs Placebo (Active Comparator): Single Ascending Dose (SAD)
  Interventions: Drug: APNmAb005; Drug: Placebo
- APNmAb005 (10 mg/kg) vs Placebo (Active Comparator): Single Ascending Dose (SAD)
  Interventions: Drug: APNmAb005; Drug: Placebo
- APNmAb005 (25 mg/kg) vs Placebo (Active Comparator): Single Ascending Dose (SAD)
  Interventions: Drug: APNmAb005; Drug: Placebo
- APNmAb005 (50 mg/kg) vs Placebo (Active Comparator): Single Ascending Dose (SAD)
  Interventions: Drug: APNmAb005; Drug: Placebo
- APNmAb005 (70 mg/kg) vs Placebo (Active Comparator): Single Ascending Dose (SAD)
  Interventions: Drug: APNmAb005; Drug: Placebo

INTERVENTIONS:
Drug: APNmAb005 — Administered by IV infusion
Drug: Placebo — Administered by IV infusion

SUMMARY:
This is a Phase 1, first-in-human (FIH), double-blinded, placebo-controlled study where healthy subjects are randomly allocated to receive APNmAb005 or placebo. Approximately 5 dosing groups (cohorts) are planned with 8 subjects (randomized to 6 active: 2 placebo) per cohort. the starting dose of APNmAb005 is 5 mg/kg and the anticipated doses for subsequent cohorts are 10, 25, 50 and 70 mg/kg. A Safety Review Team (SRT) will review data on an ongoing basis throughout the study and before progression to the next dose level cohort.

Subjects will receive a single dose of either APNmAb005 or placebo administered as a single IV infusion on Day 1 of the study and will remain in the study center until Day 3 (48 hours after dosing). They will return to the study center for 7 outpatient visits. The duration of the study, excluding screening, is approximately 71 days.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18.5 to 32 kg/m² inclusive, at screening.
* Female subjects of childbearing potential must use an acceptable method of birth control from screening until at least 90 days after study drug dosing; OR be surgically sterile; OR be postmenopausal. All female subjects must have a negative pregnancy test at screening and before the first dose of the study drug. Female subjects must also agree to refrain from egg donation during the study and for at least 90 days after study drug dosing.
* Male subjects must agree to use a condom when sexually active with a female partner of childbearing potential during the study and for at least 90 days after study drug dosing (or be surgically sterile); OR agree to practice abstinence during the study and for at least 90 days after study drug dosing. Male subjects must also agree to refrain from sperm donation during the study and for at least 90 days after study drug dosing.
* Agree to comply with all protocol requirements.
* Provide written informed consent.

Exclusion Criteria:

* Unable or unwilling to undergo venipuncture or tolerate venous access, or is unable or unwilling to undergo lumbar puncture.
* Has any significant acute or chronic medical illness that would impact the subject's ability to complete all study requirements or impact assessment of study data; or subject as had a clinically significant illness within 30 days prior to study drug dosing.
* Any medical condition or documented history that is a contraindication to lumbar puncture (e.g. bleeding disorder, spinal deformity).
* Positive COVID-19 molecular diagnostic test result at screening or prior to study drug dosing; or subject has known or suspected consequence from prior COVID-19 infection.
* History of cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal or oncogenic (with the exception of resected skin basal cell carcinoma) disease within 5 years prior to screening).

NOTE: Subjects with treated stable psychiatric conditions (e.g. anxiety, depression) are not allowed.

* Clinically significant neurological or psychiatric disorder.
* Major surgery, as determined by investigator, within 4 weeks prior to study drug dosing.
* Systolic blood pressure >140 mm Hg and/or diastolic blood pressure >90 mm Hg.
* Received any vaccine or used any prescription or over-the-counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days prior to study drug dosing.
* Consumed caffeine- or xanthine-containing products within 48 hours prior to study drug dosing.
* Subject is a smoker or has regularly used nicotine or nicotine-containing products (e.g. snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 3 months prior to study drug dosing.
* Subject is involved in vigorous or strenuous physical activity or contact sports within 24 hours prior to study drug dosing.
* Subject has donated blood or blood products >450 mL within 3 months prior to study drug dosing.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events (AEs) | Day 70
  Defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Data collected by subject observations and data collected on AE page of electronic Case Report Form (eCRF), or other documents relevant to subject safety.
Number of subjects with Treatment-emergent AEs (TEAEs) | Day 70
  Defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure. Data collected by subject observations and data collected on AE page of electronic Case Report Form (eCRF), or other documents relevant to subject safety.
Number of subjects with Serious Adverse Events (SAEs) | Day 70
  Defined as any AE for which there is a reasonable possibility that the study drug caused the AE. Data collected by subject observations and data collected on AE page of electronic Case Report Form (eCRF), or other documents relevant to subject safety.
Number of subjects with AEs resulting in Study Discontinuation | Day 70
  Data collected by subject observations and data collected on AE page of electronic Case Report Form (eCRF), or other documents relevant to subject safety.
Number of participants with Vital Sign Abnormalities | Day 70
  Measured by systolic and diastolic blood pressures, pulse rate, respiratory rate and body temperature.
Number of participants with Electrocardiogram (ECG) Abnormalities | Day 70
  Measured by 12-lead ECG
Number of participants with Clinical Laboratory Abnormalities | Day 70
  Measured by hematology, coagulation, serum chemistry and urinalysis.

SECONDARY OUTCOMES:
AUC0-t of APNmAb005 in plasma | Thru Day 70
  Area under the curve from time zero to last quantifiable concentration of APNmAb005. Measured by blood sample analysis.
AUC0-t of APNmAb005 in CSF | Thru Day 14
  Area under the curve from time zero to last quantifiable concentration of APNmAb005. Measured by cerebrospinal fluid (CSF) sample analysis.
Cmax of APNmAb005 in blood | Thru Day 70
  Maximum observed plasma concentration of APNmAb005. Measured by blood sample analysis
Cmax of APNmAb005 in CSF | Thru Day 14
  Maximum observed plasma concentration of APNmAb005. Measured by cerebrospinal fluid (CSF) sample analysis.
Tmax of APNmAb005 in blood | Thru Day 70
  Time to maximum observed plasma concentration following APNmAb005 administration. Measured by blood sample analysis
Tmax of APNmAb005 in CSF | Thru Day 14
  Time to maximum observed plasma concentration following APNmAb005 administration. Measured by cerebrospinal fluid (CSF) sample analysis.
t1/2 of APNmAb005 in plasma | Thru Day 70
  Terminal phase half-life of APNmAb005. Measured by blood sample analysis
t1/2 of APNmAb005 in CSF | Thru Day 14
  Terminal phase half-life of APNmAb005. Measured by cerebrospinal fluid (CSF) sample analysis
CL of APNmAb005 in blood. | Thru Day 70
  Total body clearance of APNmAb005 from plasma. Measured by blood sample analysis
CL of APNmAb005 in CSF | Thru Day 14
  Total body clearance of APNmAb005 from plasma. Measured by cerebrospinal fluid (CSF) sample analysis
Vd of APNmAb005 in plasma | Thru Day 70
  Volume of distribution of APNmAb005. Measured by blood sample analysis
Vd of APNmAb005 in CSF | Thru Day 14
  Volume of distribution of APNmAb005. Measured by cerebrospinal fluid (CSF) sample analysis
Number of participants with ADA formation against APNmAb005 | Thru Day 70
  Anti-drug antibody (ADA) presence measured by blood sample analysis
Number of participants with no ADA formation against APNmAb005 | Thru Day 70
  Anti-drug antibody (ADA) presence measured by blood sample analysis
Mean Total tau concentration in plasma | Thru Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean change in Total tau concentration in plasma | Baseline and Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean Total tau concentration in CSF | Thru Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis
Mean change in Total tau concentration in CSF | Baseline and Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis
Mean p-tau 181 concentration in plasma | Thru Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean change in p-tau 181 concentration in plasma | Baseline and Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean p-tau 181 concentration in CSF | Thru Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis
Mean change in p-tau 181 concentration in CSF | Baseline and Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis
Mean p-tau 217 concentration in plasma | Thru Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean change in p-tau 217 concentration in plasma | Baseline and Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean p-tau 217 concentration in CSF | Thru Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis
Mean change in p-tau 217 concentration in CSF | Baseline and Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis
Mean p-tau 231 concentration in plasma | Thru Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean change in p-tau 231 concentration in plasma | Baseline and Day 70
  Pharmacodynamic biomarker concentration measured by blood sample analysis
Mean p-tau 231 concentration in CSF | Thru Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis
Mean change in p-tau 231 concentration in CSF | Baseline and Day 14
  Pharmacodynamic biomarker concentration measured by CSF analysis

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, DO, Principal Investigator — Collaborative Neuroscience Research, LLC
Locations (1):
- Collaborative Neuroscience Research, LLC., 2600 Redondo Ave., Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No